CLINICAL TRIAL: NCT00981305
Title: Impact of Lactate-containing Vaginal Lubricant on Sexual Dysfunction in Young Breast Cancer Survivors: Prospective Randomized Controlled Trial
Brief Title: Impact of Lactate-Containing Vaginal Lubricant on Sexual Dysfunction in Young Breast Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Medical Research Collaborating Center, Seoul, Korea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNUH 0905-037-281
Record Dates: First submitted 2009-09-20; First posted 2009-09-22 (Estimated); Results first posted 2017-01-26 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2016-10

CONDITIONS: Sexual Dysfunction; Breast Cancer Survivors
Keywords: dyspareunia; breast cancer; sexual dysfunction; vaginal lubricant
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Dyspareunia; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactate-containing Vaginal Lubricant (Experimental): apply 3cc of lactate-containing vaginal lubricant before sexual intercourse or sleeping for 8wks (at least 3 times per week)
  Interventions: Drug: Lactate-containing vaginal lubricant
- Placebo (Placebo Comparator): apply 3cc of placebo vaginal lubricant before sexual intercourse or sleeping for 8wks (at least 3 times per week)
  Interventions: Drug: Placebo vaginal lubricant

INTERVENTIONS:
Drug: Lactate-containing vaginal lubricant — vaginal applying at least 3cc of lactate-containing lubricant at the time of sexual intercourse or before sleeping for 8 weeks (at least 3 times/week)
  Other Names: Clino-san(commercial name in Korea)
  Arms: Lactate-containing Vaginal Lubricant
Drug: Placebo vaginal lubricant — vaginal applying at least 3cc of placebo lubricant at the time of sexual intercourse or before sleeping for 8 weeks (at least 3 times/week)
  Other Names: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether lactate-containing vaginal lubricant is effective in the treatment of young breast cancer survivors with sexual dysfunction.

DETAILED DESCRIPTION:
Study scheme

* study arm: apply lactate-containing lubricants at the time of sexual intercourse and before sleep at least 3 times per a week for 8 weeks
* control arm: placebo apply

Outcome measures

* Female Sexual function Index (FSFI-20): at 0 wk and at 8 wk
* vaginal maturation index: at 0 wk and 8 wk
* vaginal pH: at 0 wk and 8 wk

ELIGIBILITY:
Inclusion Criteria:

* breast cancer survivors over 20 years-old
* premenopausal at the time of diagnosis
* treated with operation and chemotherapy
* newly developed dyspareunia after cancer treatment

Exclusion Criteria:

* recent (< 2 months) start or cessation of hormonal treatment (tamoxifen etc.)
* depression or other psychological problems
* active vaginal infection
* evidence of cancer recurrence
* previously use of lactate-containing lubricants
* other chronic diseases which severely disturb the sexual life

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2009-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myung Jae Jeon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Myung Jae, Jeon, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YH, Park S, Lee M, Hahn S, Jeon MJ. Effect of a pH-Balanced Vaginal Gel on Dyspareunia and Sexual Function in Breast Cancer Survivors Who Were Premenopausal at Diagnosis: A Randomized Controlled Trial. Obstet Gynecol. 2017 May;129(5):870-876. doi: 10.1097/AOG.0000000000001988. PMID 28383379

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo
Started | 69 | 67
Completed | 50 | 57
Not Completed | 19 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo | Total
Number analyzed (Participants) | 50 | 57 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (6.0) | 49.0 (5.2) | 48.8 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 57 | 107
  Male | 0 | 0 | 0
Parity [Median (Full Range); unit: pregnancies] | 2 [0 to 3] | 2 [0 to 5] | 2 [0 to 5]
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (2.4) | 23.3 (3.3) | 23.2 (2.9)
Menopause [Number; unit: participants]
  Yes | 35 | 41 | 76
  No | 15 | 16 | 31
Tamoxifen treatment [Number; unit: participants]
  Yes | 33 | 40 | 73
  No | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Change of Pain Score of Female Sexual Function Index
Description: The Female Sexual Function Index (FSFI) is a 19-item self-reported instrument used for assessing key dimensions of female sexual function over the past 4 weeks with a total of six domains being analyzed. Each of the six specific domains (desire, arousal, lubrication, orgasm, satisfaction, and pain) analyzed in the FSFI is scored on a scale ranging from 1.2 to 6.0 (desire), 0 to 6.0 (arousal, lubrication, orgasm, and pain) or 0.8 to 6.0 (satisfaction), with higher scores indicating better performance. The total score, falling in a possible range from 2.0 to 36.0, is obtained by adding the six domain scores together.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo
Number analyzed (Participants) | 50 | 57
units on a scale | 1.15 (1.59) | 1.05 (1.54)

2. Secondary Outcome: Change of a Total and Other Five Domains of Female Sexual Function Index Score
Description: as for outcome 1
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo
Number analyzed (Participants) | 50 | 57
units on a scale
  Total | 2.85 (4.10) | 3.81 (5.10)
  Desire | 0.19 (1.03) | 0.45 (0.86)
  Arousal | 0.42 (0.72) | 0.45 (0.90)
  Lubrication | 0.59 (1.23) | 0.77 (1.50)
  Orgasm | 0.38 (0.81) | 0.67 (0.94)
  Satisfaction | 0.11 (0.83) | 0.43 (1.06)

3. Secondary Outcome: Change of Vaginal pH
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo
Number analyzed (Participants) | 50 | 57
pH | -0.75 (0.52) | -0.02 (0.59)

4. Secondary Outcome: Change of Vaginal Maturation Index
Description: Vaginal maturation index is a ratio obtained by performing a random cell count of the three major cell types shed from the vaginal squamous epithelium: parabasal, intermediate, and superficial cells. The higher the maturation index, the higher the number of mature cells (those designated superficial and intermediate).
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: vaginal maturation index
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo
Number analyzed (Participants) | 50 | 57
vaginal maturation index | 4.73 (10.37) | 1.00 (8.50)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Lactate-containing Vaginal Lubricant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/57
Other Adverse Events (participants affected / at risk) | 7/50 | 7/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lactate-containing Vaginal Lubricant (N=50) | Placebo (N=57)
Vaginal itching (Reproductive system and breast disorders) | 5 | 5
Vaginal irritation (Reproductive system and breast disorders) | 0 | 1
Both (Reproductive system and breast disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No